CLINICAL TRIAL: NCT06115343
Title: Consciousness in Adolescents The Effect of Awareness Practice on Self-Efficacy and Risky Behaviors
Brief Title: Conscious Awareness Practice in Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Yunus Omer Arık, Teacher, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MINDFULNESS PRACTICE
Record Dates: First submitted 2023-10-29; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Risky Behavior
Keywords: Conscious Awareness; Self-Efficacy; adolescent
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Conscious Awareness application consists of 6 recordings of 30 minutes for 6 weeks.
  Interventions: Behavioral: Mindfulness
- Control Group (No Intervention): Participants in the control group engage in 6 sessions of 30-minute social activity for 6 weeks.

INTERVENTIONS:
Behavioral: Mindfulness — Conscious awareness practice was carried out in 6 sessions. Various inventories are used depending on the nature of the session. For example, in the leaf theme, participants are asked to close their eyes and put their thoughts from the past on a leaf and drop them into running water.
  Arms: Experimental Group

SUMMARY:
The aim of this study is to reveal the effect of mindfulness on self-efficacy and risky behaviors in adolescents.

DETAILED DESCRIPTION:
This randomized controlled experimental study was carried out between 18 September and 27 October at Istanbul Bağcılar Necmettin Erbakan Science High School with a total of 60 students (30 experimental group / 30 control group). Research data were collected from the Conscious Awareness-Based Self-Efficacy Scale-Revised (BFÖS-Y), Risky Behaviors Scale (RDS) and Personal Information Form. Ethics committee approval, written institutional permission and written permission from the participants were obtained for the research. In the first week, pre-tests were given to the experimental and control groups, and the experimental group was given 30 minutes of mindfulness training. Mindfulness training continued to be given to the experimental group for the next 5 weeks, and post-tests were given to the experimental and control groups in the last week.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 14 and 18
* Agree to participate in the study
* Being literate and speaking Turkish fluently
* Have communication and understanding skills

Exclusion Criteria:

* Having a physical health problem that may impair group cohesion and integrity

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-11-20 (Estimated)

PRIMARY OUTCOMES:
Change in The Effect of Mindfulness Training on Self-Efficacy in Adolescents. | [Time Frame: up to 6 weeks]
  Mindfulness-Based Self-Efficacy Scale scores range from 22 to 110. 22 is the lowest possible score and 110 is the highest possible score. The scale consists of 22 items and 6 dimensions. A low score indicates that their conscious-awareness-based self-efficacy is weak.
Change in The Impact of The Functioning of Detention Education in Adolescents. | [Time Frame: up to 6 weeks]
  Risk Behavior Scale scores range from 36 to 180. 36 is the lowest possible score and 180 is the highest possible score. The scale consists of 36 items and 6 dimensions. Getting a high score from the scale indicates the intensity of risky behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Yunus Ömer ARIK, Teacher, Principal Investigator — pskdan.yunusomerarik@gmail.com
Locations (1):
- Korkut Ata University, Osmaniye, Center, Turkey (Türkiye)